CLINICAL TRIAL: NCT05845736
Title: The Impact of Dementia and Neurocognitive Disorders on Hypertension Treatment in the Very Elderly: the TAHOC Study
Brief Title: The Impact of Dementia and Neurocognitive Disorders on Hypertension Treatment in the Elderly
Acronym: TAHOC
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pr Athanase BENETOS, principal investigator, Central Hospital, Nancy, France
Other Study IDs: 2023PI017
Record Dates: First submitted 2023-03-26; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Neurocognitive Disorders; Dementia; Hypertension; Aged, 80 and Over
Keywords: Neurocognitive Disorders; Dementia; Hypertension; Aged, 80 and over
MeSH Terms: conditions — Neurocognitive Disorders; Dementia; Hypertension | interventions — Antihypertensive Agents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- control group: absence of neurocognitive disorder (ND), Mini-Mental State Examination (MMSE) from 27 to 30 inclusive
  Interventions: Drug: Antihypertensive Agents
- mild neurocognitive disorder: MMSE from 21 to 26 inclusive
  Interventions: Drug: Antihypertensive Agents
- moderate neurocognitive disorder: MMSE from 11 to 20 inclusive
  Interventions: Drug: Antihypertensive Agents
- severe neurocognitive disorder: MMSE less than or equal to 10
  Interventions: Drug: Antihypertensive Agents

INTERVENTIONS:
Drug: Antihypertensive Agents — number of hypertensive drugs

SUMMARY:
Neurocognitive disorders and hypertension occur commonly with aging. While, by definition, older adults are at high cardiovascular risk, there is no guideline exist currently on blood pressure management of elderly hypertension. However, studies have shown that in aging adults, high blood pressure helps prevent against cognitive decline, and low blood pressure on antihypertensive drugs could accelerate it. This study aims at investigating if pharmacological treatment of hypertension in the very elderly is influenced by presence and severity of neurocognitive disorders. Our research hypothesis is that the drug management of hypertension in patients 80 years of age or older more is all the less aggressive as the neurocognitive disorders are advanced.

ELIGIBILITY:
Inclusion Criteria:

* to be 80 years of age
* with history of hypertension and/or on hypertensive drug(s)

Exclusion Criteria:

* legal protection measure.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients aged 80 years or more and hypertensive who received a Comprehensive Geriatric Assessment (including a mini mental state examination) as part of a frailty, memory or oncogeriatric assessment, in day hospital in the geriatric department in University Hospital of Nancy in 2022.
Sampling Method: Non-Probability Sample
Enrollment: 353 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
number of antihypertensive agents | during inclusion
  among ACEI/ARB2, calcium channel blocker, thiazides and related, central antihypertensive beta blocker

SECONDARY OUTCOMES:
class of antihypertensive medications | during inclusion
  among ACEI/ARB2, calcium channel blocker, thiazides and related, central antihypertensive beta blocker
systolic and diastolic blood pressure | during inclusion
  blood pressure measured with upper arm cuffs
orthostatic hypotension | during inclusion
  a systolic blood pressure decrease of at least 20 mm Hg or a diastolic blood pressure decrease of at least 10 mm Hg within three minutes of standing

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Régional Universitaire de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided